CLINICAL TRIAL: NCT07213557
Title: Randomized Phase 2 Study of Simvastatin in Patients With ARID1A Mutated Advanced Gastrooesophageal Carcinoma Treated With Nivolumab and Oxaliplatin- Based Chemotherapy as First-line Treatment (The ARES Trial)
Brief Title: Simvastatin Efficacy in ARID1A Mutated Advanced gastroESophageal Carcinoma Treated With Immunotherapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARES; 2024-519591-39-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-22; First posted 2025-10-09 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-09

CONDITIONS: Advanced or Metastatic Gastrooesophageal Carcinoma
Keywords: HER2 negative; ARID1A mutated; Simvastatin; gastrooesophageal carcinoma; liquid biopsy
MeSH Terms: interventions — Simvastatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ARM A - standard (Active Comparator): Patients with HER2 negative aGEC eligible for the standard treatment with nivolumab and oxaliplatin- based chemotherapy (CPS ≥ 5) will be evaluated for ARID1A expression by immunohistochemistry on tumor tissue. Patients with ARID1A mutated will be randomized to receive standard nivolumab and oxaliplatin- based chemotherapy (standard arm, ARM A) or simvastatin in combination with standard nivolumab and oxaliplatin-based chemotherapy (experimental arm, ARM B)
  Interventions: Drug: standard nivolumab and oxaliplatin- based chemotherapy
- ARM B (Experimental): Patients with HER2 negative aGEC eligible for the standard treatment with nivolumab and oxaliplatin- based chemotherapy (CPS ≥ 5) will be evaluated for ARID1A expression by immunohistochemistry on tumor tissue. Patients with ARID1A mutated will be randomized to receive standard nivolumab and oxaliplatin- based chemotherapy (standard arm, ARM A) or simvastatin in combination with standard nivolumab and oxaliplatin-based chemotherapy (experimental arm, ARM B)
  Interventions: Drug: simvastatin in combination with standard nivolumab and oxaliplatin-based chemotherapy
- ARM C (Other): Observational Cohort: patients with ARID1A not mutated of observational cohort (ARM C) will be treated with standard treatment with nivolumab and oxaliplatin-based chemotherapy and compared with standard ARM A as exploratory comparison to evaluate the predictive value for immunotherapy of ARID1A.
  Interventions: Drug: standard nivolumab and oxaliplatin- based chemotherapy

INTERVENTIONS:
Drug: standard nivolumab and oxaliplatin- based chemotherapy — Nivolumab will be administered as 30 minutes intravenous infusion at the dosage of 360 mg every 3 weeks or 240 mg every 2 weeks as flat dose followed by investigator's choice of oxaliplatin-based chemotherapy regimen:
  * XELOX (oxaliplatin 130 mg/m2 on day 1 and capecitabine 1,000 mg/m2 orally twice daily on days 1- 14 administered every 3 weeks) or
  * mFOLFOX6 (oxaliplatin 85 mg/m2 on day 1 followed by lederfolin 200 mg m2 on day 1, fluorouracil 400 mg m2 on day 1 and 2,400 mg m2 continuous infusion over 46 hours every 2 weeks)
  Arms: ARM A - standard; ARM C
Drug: simvastatin in combination with standard nivolumab and oxaliplatin-based chemotherapy — Nivolumab will be administered as 30 minutes intravenous infusion at the dosage of 360 mg every 3 weeks or 240 mg every 2 weeks as flat dose followed by investigator's choice of oxaliplatin-based chemotherapy regimen:
  * XELOX (oxaliplatin 130 mg/m2 on day 1 and capecitabine 1,000 mg/m2 orally twice daily on days 1- 14 administered every 3 weeks) or
  * mFOLFOX6 (oxaliplatin 85 mg/m2 on day 1 followed by lederfolin 200 mg m2 on day 1, fluorouracil 400 mg m2 on day 1 and 2,400 mg m2 continuous infusion over 46 hours every 2 weeks)
  * SIM will be administered per os daily at a fixed dosage of 40 mg that represents the recommended dose as cholesterol lowering agents.
  Arms: ARM B

SUMMARY:
The investigators hypothesize that simvastatin (SIM) may improve the efficacy of first- line Nivolumab and Oxaliplatin-based chemotherapy, extending progression-free survival (PFS) as compared with Nivolumab and chemotherapy alone in patients with HER2 negative and ARID1A mutated advanced gastrooesophageal carcinoma (aGEC).

Correlative mechanistic studies on tissue and blood samples, could help understanding the evolutionary dynamics of tumors in response to therapy thus optimizing the treatment approach and adding new insight into the antitumor mechanism of the combination approach.

DETAILED DESCRIPTION:
This study is a multicentric open label academic non comparative randomized phase-2 study.

Before starting study treatment, at the time of enrollment, patients, with aGEC HER2 negative with ARID1A mutation in tumors candidates for immunotherapy (CPS ≥ 5), will be randomized electronically 1:1 to one of the two arms:

* ARM A, standard treatment with nivolumab + oxaliplatin- based chemotherapy (mFOLFOX6 or XELOX regimen)
* ARM B, experimental treatment with simvastatin oral daily at a fixed dosage of 40 mg, in addition to standard treatment with nivolumab + oxaliplatin-based chemotherapy (mFOLFOX6 or XELOX regimen).

Nivolumab will be administered as flat dose of 360 mg every 3 weeks or 240 mg every 2 weeks with investigator's choice of oxaliplatin-based chemotherapy regimen:

* XELOX (oxaliplatin 130 mg/m2 on day 1 and capecitabine 1,000 mg/m2 orally twice daily on days 1-14 administered every 3 weeks) or
* mFOLFOX6 (oxaliplatin 85 mg/m2 on day 1 followed by lederfolin 200 mg m2 on day 1, fluorouracil 400 mg m2 on day 1 and 2,400 mg m2 continuous infusion over 46 hours every 2 weeks) Patients will continue to receive study treatment until treatment failure as previous defined, unacceptable toxicity, physician's decision, patient's refusal, or any other discontinuation criteria.

Patients who are progression free after 8 cycles (24 weeks) of XELOX or 12 cycles (24 weeks) of mFOLFOX6 treatment will continue maintenance with fluorouracile (lederfolin 200 mg m2 on day 1, fluorouracil 400 mg m2 on day 1 and 2,400 mg m2 continuous infusion over 46 hours every 2 weeks) or capecitabine (capecitabine 1,250 mg/m2 orally twice daily on days 1-14 administered every 3 weeks), as previously assigned until treatment failure as reported above.

28 aGEC HER2 negative and ARID1A mutated patients will be required along to other 28 aGEC HER2 negative and ARID1A mutated patients as calibration arm, for a total of 56 subjects.

All subjects who finish treatment, whichever the reason, will enter in the follow-up. All patients will be followed until death and data on subsequent treatment will be collected.

An initial safety run-in phase involves a safety evaluation after the first 6 patients are randomly assigned to Arm B. Enrollment will be paused after the first 6 patients randomly assigned to Arm B complete 2 cycles of treatment. The enrollment will be interrupted if the treatment combination will be judged not feasible and major safety concerns will arise. A safety review will be conducted, and recommendations will be made by the Steering Committee. The study will continue if there are 2 or fewer adverse events (AEs) of grade 3 or higher deemed related to the addition of simvastatin to the standard treatment with nivolumab + oxaliplatin-based chemotherapy.

All measurable and non-measurable lesions must be documented at screening (within 28 days prior to randomization) and re-assessed at each subsequent tumor evaluation (every 12 weeks). Tumor assessment by CT scan (chest, abdomen and pelvis) or MRI (abdomen and pelvis); CEA, CA 19.9; and any other tests resulted positive during baseline staging, will be performed every 12 weeks during treatment until treatment failure in both arms. Patients discontinuing study treatment without progressive disease, will undergo tumor assessments every 12 weeks until progressive disease or study withdrawal.

Toxicities will be evaluated at each clinical visit throughout the study treatment and up to 4 weeks after last cycle of treatment accordingly to the Common Terminology Criteria for Adverse Events (AEs) of the National Cancer Institute (CTCAE-NCI) version 5.0.

Quality of Life will be assessed by the EORTC QLQ-C30 v.3.0 questionnaire that will be completed by patients at baseline (prior to treatment, once eligibility is confirmed) and every 12 weeks until disease progression or, treatment failure.

HER2-negative aGEC patients with ARID1A non mutated tumors of observational cohort who are candidates for immunotherapy (ARM C) will be treated with standard treatment with nivolumab and oxaliplatin-based chemotherapy in the same way as the patients in ARM A (28 patients)

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent to study procedures and to correlative studies.
2. Aged ≥ 18.
3. Histologically proven of gastrooesophageal carcinoma
4. Diagnosis of advanced not operable or metastatic disease.
5. HER2 negative and ARID1A mutated status at initial diagnosis.
6. Available tumor tissue sample.
7. No prior treatments (chemotherapy, radiation or surgery) for aGEC. Surgery for primary GEC tumor before starting treatment is allowed.
8. Patient candidate to standard treatment with nivolumab and oxaliplatin-based chemotherapy as clinical practice (combined positive score ≥ 5).
9. Eastern Cooperative Oncology Group (ECOG) Performance Status

   ≤ 1 at study entry.
10. Imaging-documented measurable disease, according to RECIST 1.1 criteria.
11. Estimated life expectancy of more than 12 weeks.
12. Adequate bone marrow hematological function: absolute neutrophil count (ANC) ≥ 1.5 x 109/L and platelet count ≥ 100 x 109/L and hemoglobin ≥ 9 g/dL.
13. Adequate liver function: total bilirubin ≤ 1.5 x upper limit of normal (ULN) or ≤ 2 (in case of biliary stent) and aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 5 X ULN.
14. Adequate renal function: serum creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 60 mL/min in males and ≥50 mL/min in females (calculated according to Cockroft-Gault formula).
15. Known dihydropyrimidine dehydrogenase (DPYD) activity is mandatory. The same criteria, except for the status of ARID1A, will be followed to select the 28 consecutive HER2-negative and ARID1A non mutated aGEC patients of observational cohort.

Exclusion Criteria:

1. Prior malignancy within five years. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
2. Prior chemotherapy or any other medical treatment for aGEC (previous adjuvant chemotherapy is allowed if terminated > 12 months previously).
3. Any contraindication to Nivolumab, simvastatin or oxaliplatin-based chemotherapy.
4. Patients who have treatment with statins or fibrates or any medication for hypercholesterolemia.
5. Major surgical intervention within 4 weeks prior to enrollment.
6. Pregnancy and breast-feeding.
7. Any brain metastasis.
8. Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the investigator's opinion makes it undesirable for the patient to participate in the study, or which would jeopardize compliance with the protocol, or would interfere with the results of the study.
9. History of poor co-operation, non-compliance with medical treatment, unreliability or any condition that may impair the patient's understanding of the Informed consent form.
10. Participation in any interventional drug or medical device study within 30 days prior to treatment start.
11. Sexually active males and females (of childbearing potential) unwilling to practice contraception (barrier contraceptive measure or oral contraception) during the study and until 6 months after the last trial treatment.
12. Hypesensitivity to simvastatin.
13. Acute hepatitis or chronic hepatitis.
14. Personal or familial anamnesis of severe hepatopathy.
15. Known coagulation disorders. The same criteria will be followed to select the 28 consecutive HER2-negative and ARID1A non mutated aGEC patients of observational cohort.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival rate at 1-year (PFS 1-year) | up to 1 year to randomization
  Progression Free Survival rate at 1-year (PFS 1-year) PFS 1-year is defined as the rate of assessable patients alive and not progressed after 1 year from initiation of study (i.e randomization) to the first documentation of: objective disease progression by RECIST 1.1 criteria, including deterioration of clinical conditions preventing radiological restaging, treatment interruption due to AEs followed by initiation of an alternative antineoplastic treatment, or death due to any cause, whichever occurs first in one year. It will be measured as the rate of assessable patients alive and without disease progression, as previously defined, at 1 year.

SECONDARY OUTCOMES:
Objective Tumor Response Rate (ORR) | up to 1 year last patients randomized
  Objective Tumor Response Rate (ORR) defined as the proportion of patients with complete/partial response, assessed according to RECIST criteria 1.1.
Disease Control Rate (DCR) | up to 1 year to randomization
  Disease Control Rate (DCR) defined as the proportion of patients with complete/partial response and stable disease as their best response, assessed according to RECIST criteria 1.1.
Progression-free survival (PFS) | up to 1 year to randomization
  Progression-free survival (PFS) measured as the time from the date of randomization until the date of the first observation of disease progression or death due to any cause, whichever occurs first, or the last date of follow up.
Overall survival (OS) | up to 1 year to randomization
  Overall survival (OS) calculated as the time from the date of randomization until the date of death from any cause, or the last date of follow up.
Safety evaluated as adverse events graded according to NCI CTCAE v 5.0. | From the start of the first treatment cycle until the end of active treatment
  Safety evaluated as adverse events graded according to NCI CTCAE v 5.0.
Quality of life (QoL) | at baseline and every 12 weeks until disease progression.
  Quality of life (QoL) investigated through the EORTC QLQ-C30